CLINICAL TRIAL: NCT00363168
Title: Ranibizumab in Hemorrhagic Choroidal Neovascularization Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Neil M. Bressler, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00001650
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-09

CONDITIONS: Choroidal Neovascularization
Keywords: Hemorrhagic Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 0.3 mg/0.05 ml dose of ranibizumab
  Interventions: Drug: Ranibizumab
- B (Experimental): 0.5 mg/0.05 ml dose of ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.3 mg/0.05 ml dose
  Other Names: Lucentis
  Arms: A
Drug: Ranibizumab — 0.5 mg/0.05 ml dose
  Other Names: Lucentis
  Arms: B

SUMMARY:
This research is being done to look at the effects of an experimental drug, ranibizumab, on a condition called "predominantly hemorrhagic subfoveal choroidal neovascularization (CNV)" due to wet age-related macular degeneration.

A predominantly hemorrhagic CNV lesion is diagnosed when at least 50% of the choroidal neovascular lesion is occupied by blood under the retina. We want to find out if injections of ranibizumab into the eye will help patients with this condition.

DETAILED DESCRIPTION:
This study is a randomized, interventional case series. A total of 10 patients, seen in the Retina Division of the Wilmer Eye Institute, will be enrolled. Subjects will be randomized to either 0.3 mg or 0.5 mg intravitreal injections of ranibizumab, which will be performed monthly for 3 doses. Further monthly injections are at the discretion of the examiner, and may be withheld if there is lack of continued improvement (defined as lack of improvement of at least 5 letters on an eye chart compared with 2 previous consecutive visits or lack of decrease of the retinal center point thickness of at least 50 microns compared with 2 previous consecutive visits) or complete success (defined as visual acuity of 20/20 or better or retinal center point thickness <225 microns).

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Predominantly hemorrhagic subfoveal CNV (at least 50% of the lesion composed of hemorrhage) from age-related macular degeneration (AMD) resulting in visual acuity of 20/40 or worse.
* Age greater than 50 years.
* Participant must have media clear enough to permit fundus photography, fluorescein angiography, and optical coherence tomography.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Known hypersensitivity to humanized monoclonal antibodies
* History (within past 6 months) or evidence of severe cardiac disease (apparent in electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within 6 months prior to baseline, atrial or ventricular tachyarrhythmias requiring ongoing treatment).
* History of stroke within 6 months of study entry.
* Current acute ocular or periocular infection.
* Any major surgical procedure within one month of study entry.
* Known serious allergies to fluorescein dye.
* Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, Protein Kinase C inhibitors, etc) within last 6 months.
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye within the last 6 months.
* History of subfoveal laser treatment in the study eye.
* History of other visually-limiting conditions such as optic neuropathy, amblyopia, choroidal neovascularization due to causes other than AMD in the study eye.
* Ocular inflammation (including trace or above) in the study eye.
* Inability to comply with study or follow up procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil M. Bressler, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Chang MA, Do DV, Bressler SB, Cassard SD, Gower EW, Bressler NM. Prospective one-year study of ranibizumab for predominantly hemorrhagic choroidal neovascular lesions in age-related macular degeneration. Retina. 2010 Sep;30(8):1171-6. doi: 10.1097/IAE.0b013e3181dd6d8a. PMID 20827138

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab Dose A: 0.3 mg/0.05 ml intravitreal injection
- Ranibizumab Dose B: 0.5 mg/0.05 ml intravitreal injection
Period: Overall Study
Arm/Group | Ranibizumab Dose A | Ranibizumab Dose B
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Dose A | Ranibizumab Dose B | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Avoiding 15 or More Letter Loss of Best Corrected Visual Acuity From Baseline to 12 Months on an Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Chart Measured at 4 Meters.
Description: Visual acuity measured prior to first treatment with ranibizumab and at 12 months following the first treatment were compared for each subject enrolled in the study. The 12 month follow-up visual acuity was subtracted from the baseline visual acuity. Avoiding a 15 or more letter loss in visual acuity was considered a successful outcome.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Ranibizumab Dose A | Ranibizumab Dose B
Number analyzed (Participants) | 5 | 2
participants | 5 | 2

2. Secondary Outcome: Retinal Changes on Funduscopy
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Retinal Thickness Measured by Optical Coherence Tomography (OCT)
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Fluorescein Leakage on Fluorescein Angiography
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Number of Subjects Experiencing Complications Related to Drug or Its Administration
Description: Potential complications included:
  * Deterioration of best-corrected visual acuity by 3 or more lines
  * Development of intraocular inflammation
  * Development of elevated intraocular pressure
  * Development of other ocular or systemic adverse effects.
  Subjects were monitored for potential drug-related ocular adverse effects: intraocular inflammation (uveitis), endophthalmitis, central retinal vein occlusion, transient elevation of IOP, acute reduction in the visual acuity, vitreous hemorrhage, injection-site pain, retinal hemorrhage, posterior vitreous detachment, and subconjunctival hemorrhage. Subjects were monitored for potential adverse effects of intravitreal injections: crystalline lens penetration, retinal break and/or detachment, vitreous hemorrhage, inflammation, and infection. Potential systemic adverse effects were captured by monitoring vital functions such as cardiovascular function, nervous system function, renal function, and gastrointestinal function.
Time Frame: 12 months after last injection
Measure: Number; unit: participants
Arm/Group | Ranibizumab Dose A | Ranibizumab Dose B
Number analyzed (Participants) | 5 | 2
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ranibizumab Dose A | Ranibizumab Dose B
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No